CLINICAL TRIAL: NCT07002814
Title: Feasibility of Direct Oral Challenges in Private Practice Setting for the Evaluation of Mild Delayed Reactions to Beta-lactams in Children
Brief Title: Direct Oral Challenges in Private Practice Setting to Delabeling Children With Beta-lactam Allergy
Acronym: Betalactaville
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250276; ID-RBC (Other: 2025-A00658-41)
Record Dates: First submitted 2025-04-29; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Allergy
Keywords: Beta-lactams; Allerg; Allergology; Direct oral challenge
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children requiring a direct oral challenge (DOC): Children previously labeled with suspected beta-lactam allergy, requiring a direct oral challenge (DOC) to confirm or rule out true hypersensitivity

SUMMARY:
The purpose of this study is to demonstrate the feasibility of direct oral challenge performed in private practice setting for children with suspected benign delayed allergy to beta-lactams.

The results of this study could help establish recommendations for conducting direct oral challenge in primary care settings to delabeling children with benign delayed reactions to beta-lactams.

DETAILED DESCRIPTION:
Approximately 10% of children are labeled as allergic to beta-lactams (BL). Consequently, they receive alternative antibiotics with a broader spectrum but lower efficacy, leading to increased infectious morbidity and mortality, a higher risk of colonization with antibiotic-resistant bacteria, and elevated healthcare costs. However, true BL allergy is only confirmed in 5-10% of cases. Therefore, an essential challenge is to promptly identify non-allergic children to prevent unnecessary medical restrictions.

The most common reactions are delayed and benign. Current guidelines recommend evaluating these reactions through direct oral challenge (DOC) without prior allergological assessment, as traditional diagnostic methods, particularly skin tests, have poor sensitivity in this context. However, the optimal setting for conducting these tests remains debated, particularly regarding whether they can be initiated in hospital settings or private medical practices.

To date, over 8,300 DOCs have been performed in children, predominantly in hospital-based consultations. These tests have demonstrated a favorable safety profile, with positive DOC reactions often being of the same nature and less severe than the initial reported reaction. While many physicians perform DOCs in private practice, data on their use in pediatric populations remain scarce.

The primary objective of this study is to assess the feasibility of DOCs conducted in private medical practices for children with suspected benign delayed allergy to BL

ELIGIBILITY:
Inclusion Criteria:

* Population: Children's age between 0 and 17 years
* Child who has undergone a direct oral challenge in a private medical practice and a follow-up consultation within 7 to 14 days for suspected delayed allergy to amoxicillin +/- clavulanate or cefpodoxime or cefixime with the following characteristics:
* delayed reaction (onset > 1 hour after treatment start),
* mild reaction (isolated urticaria or Maculopapular exanthema),
* Absence of warning signs suggestive of a severe cutaneous adverse reaction (erythroderma, presence of bullae, vesicles, pustules, target lesions, involvement of oral, genital, or ocular mucosa, facial edema, general condition impairment, organ failure, duration > 7 days).

Exclusion Criteria:

* Informed children or holders of parental authority objecting to the use of patient data in the study.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child who underwent a direct oral challenge in a private practice setting for suspected mild delayed allergy to a beta-lactam
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of direct oral challenge (DOC) for beta-lactam allergy assessment | Day 14
  Demonstrate the feasibility of direct oral challenges (DOCs) performed in private medical practices for the evaluation of delayed and benign reactions to beta-lactams in children by collecting the amount of positive and negative DOC results and benign reactions description.

SECONDARY OUTCOMES:
Negative and positive tests reaction nature comparison | Day 14
  Collect and compare the nature of reactions between children with positive and negative direct oral challenge
Negative and positive tests reaction chronology comparison | Day 14
  Collect and compare chronology of reactions between children with positive and negative direct oral challenge.
Negative and positive tests reaction duration comparison | Day 14
  Collect and compare duration of reactions between children with positive and negative direct oral challenge.
Negative and positive tests reactions index comparison | Day 14
  Index reactions between children with positive and negative direct oral challenge.
Reactions nature in positive tests | Day 14
  Collect and analyse the nature of reactions in positive direct oral challenge
Reactions extension in positive tests | Day 14
  Collect and analyse the extension of reactions in positive direct oral challenge
Reactions duration in positive tests | Day 14
  Collect and analyse the duration of reactions in positive direct oral challenge

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien LE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castells M, Khan DA, Phillips EJ. Penicillin Allergy. N Engl J Med. 2019 Dec 12;381(24):2338-2351. doi: 10.1056/NEJMra1807761. No abstract available. PMID 31826341
- [Background] Khan DA, Banerji A, Blumenthal KG, Phillips EJ, Solensky R, White AA, Bernstein JA, Chu DK, Ellis AK, Golden DBK, Greenhawt MJ, Horner CC, Ledford D, Lieberman JA, Oppenheimer J, Rank MA, Shaker MS, Stukus DR, Wallace D, Wang J; Chief Editor(s):; Khan DA, Golden DBK, Shaker M, Stukus DR; Workgroup Contributors:; Khan DA, Banerji A, Blumenthal KG, Phillips EJ, Solensky R, White AA; Joint Task Force on Practice Parameters Reviewers:; Bernstein JA, Chu DK, Ellis AK, Golden DBK, Greenhawt MJ, Horner CC, Ledford D, Lieberman JA, Oppenheimer J, Rank MA, Shaker MS, Stukus DR, Wallace D, Wang J. Drug allergy: A 2022 practice parameter update. J Allergy Clin Immunol. 2022 Dec;150(6):1333-1393. doi: 10.1016/j.jaci.2022.08.028. Epub 2022 Sep 17. No abstract available. PMID 36122788
- [Background] Gomes ER, Brockow K, Kuyucu S, Saretta F, Mori F, Blanca-Lopez N, Ott H, Atanaskovic-Markovic M, Kidon M, Caubet JC, Terreehorst I; ENDA/EAACI Drug Allergy Interest Group. Drug hypersensitivity in children: report from the pediatric task force of the EAACI Drug Allergy Interest Group. Allergy. 2016 Feb;71(2):149-61. doi: 10.1111/all.12774. Epub 2015 Nov 17. PMID 26416157
- [Background] Sousa-Pinto B, Tarrio I, Blumenthal KG, Araujo L, Azevedo LF, Delgado L, Fonseca JA. Accuracy of penicillin allergy diagnostic tests: A systematic review and meta-analysis. J Allergy Clin Immunol. 2021 Jan;147(1):296-308. doi: 10.1016/j.jaci.2020.04.058. Epub 2020 May 21. PMID 32446963
- [Background] Srisuwatchari W, Phinyo P, Chiriac AM, Saokaew S, Kulalert P. The Safety of the Direct Drug Provocation Test in Beta-Lactam Hypersensitivity in Children: A Systematic Review and Meta-Analysis. J Allergy Clin Immunol Pract. 2023 Feb;11(2):506-518. doi: 10.1016/j.jaip.2022.11.035. Epub 2022 Dec 14. PMID 36528293
- [Background] Demoly P, Adkinson NF, Brockow K, Castells M, Chiriac AM, Greenberger PA, Khan DA, Lang DM, Park HS, Pichler W, Sanchez-Borges M, Shiohara T, Thong BY. International Consensus on drug allergy. Allergy. 2014 Apr;69(4):420-37. doi: 10.1111/all.12350. PMID 24697291
- [Background] Chow TG, Patel G, Mohammed M, Johnson D, Khan DA. Delabeling penicillin allergy in a pediatric primary care clinic. Ann Allergy Asthma Immunol. 2023 May;130(5):667-669. doi: 10.1016/j.anai.2023.01.034. Epub 2023 Feb 2. No abstract available. PMID 36738783
- [Background] Savic L, Ardern-Jones M, Avery A, Cook T, Denman S, Farooque S, Garcez T, Gold R, Jay N, Krishna MT, Leech S, McKibben S, Nasser S, Premchand N, Sandoe J, Sneddon J, Warner A. BSACI guideline for the set-up of penicillin allergy de-labelling services by non-allergists working in a hospital setting. Clin Exp Allergy. 2022 Oct;52(10):1135-1141. doi: 10.1111/cea.14217. Epub 2022 Sep 21. PMID 36128691
- [Background] Waldron JL, Hackett J, Chaung YL, Rodway P, Clark M, Trubiano JA, Chua KYL. Oral penicillin challenge in adult community practice and primary care in Australia. J Allergy Clin Immunol Pract. 2023 Dec;11(12):3786-3788.e3. doi: 10.1016/j.jaip.2023.08.013. Epub 2023 Aug 10. No abstract available. PMID 37572750
- [Background] Duong TA, Valeyrie-Allanore L, Wolkenstein P, Chosidow O. Severe cutaneous adverse reactions to drugs. Lancet. 2017 Oct 28;390(10106):1996-2011. doi: 10.1016/S0140-6736(16)30378-6. Epub 2017 May 2. PMID 28476287
- [Background] Jaoui A, Delalande D, Siouti S, Benoist G, Seve E, Ponvert C, Scheinmann P, Faour H, Neuraz A, Garcelon N, Delacourt C, Lezmi G. Safety and cost effectiveness of supervised ambulatory drug provocation tests in children with mild non-immediate reactions to beta-lactams. Allergy. 2019 Dec;74(12):2482-2484. doi: 10.1111/all.13871. Epub 2019 May 31. No abstract available. PMID 31087349